CLINICAL TRIAL: NCT01390389
Title: Exploring the Effects of Coenzyme Q10 on Bioenergetics Metabolism in Geriatric Bipolar Depression: A 31 Phosphorus MR Spectroscopy Study
Brief Title: Exploring the Effects of Coenzyme Q10 on Bioenergetics Metabolism in Geriatric Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brent Forester, PI, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-P-000980; K23MH077287 (NIH)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Bipolar Depression
Keywords: Geriatric bipolar depression; MR Spectroscopy; Coenzyme Q10; Mitochondrial Dysfunction
MeSH Terms: conditions — Bipolar Disorder; Mitochondrial Diseases | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoQ10 (Experimental): Subjects who meet DSM-IV diagnostic criteria for Bipolar Disorder, Current Episode Depressed are assigned to this arm and administered the Coenzyme Q10 intervention. CoQ10 dosing guidelines:
  * Visit 1 (Baseline) start at 400mg once a day for two weeks
  * Visit 2 (within 7 days of Baseline visit) increase to 800 mg once a day for two weeks
  The dosage of CoQ10 can be titrated in a more gradual manner depending on clinical response and tolerability of the medication, but cannot be titrated any more rapidly than the schedule above.
  Interventions: Drug: Coenzyme Q10
- Control (No Intervention): Subjects without a known psychiatric disorder and/or unstable medical illness are assigned to the control group. The control subjects are not given CoQ10.

INTERVENTIONS:
Drug: Coenzyme Q10 — Single pill consists of 400 mg and is delivered PO.
  CoQ10 dosing guidelines:
  * Visit 1 (baseline) start at 400mg once a day for two weeks
  * Visit 2 (within 7 days of baseline visit) increase to 800 mg once a day for two weeks
  The dosage of CoQ10 can be titrated in a more gradual manner depending on clinical response and tolerability of the medication, but cannot be titrated any more rapidly than the schedule above.
  Other Names: ubiquinone
  Arms: CoQ10

SUMMARY:
The investigators propose to study and compare measures of brain energy metabolism in geriatric bipolar individuals and healthy older adults. The investigators would also like to investigate changes in brain energy metabolites associated with CoQ10 administration in older bipolar individuals. Finally, resting state functional Magnetic Resonance Imaging (fMRI) will be conducted in order to explore frontal and limbic circuitry in geriatric bipolar disorder.

* Primary Hypothesis: Baseline beta NTP and NAA will be lower, and PCr and lactate higher in Geri BPD compared with older healthy controls
* Secondary Hypothesis: Changes in PCr and beta NTP will be demonstrated in Geri BD group challenged with CoQ 10.

DETAILED DESCRIPTION:
Research Design and Methods:

Bipolar Depressed Subjects:

The Bipolar Depressed group will consist of 10 subjects (for the purposes of this study we would like to be able to recruit up to 30 subjects, with the goal of getting 10 to complete the protocol), ages 55-89, meeting DSM IV-TR criteria for bipolar disorder, current episode depressed, with depression severity rated by the MADRS and the Clinical Global Impression of severity scale (CGI). The Young Mania Rating Scale (YMRS) will be used to assess concomitant manic symptoms and neuropsychological measures to assess cognitive status. Subjects with any current or previous Axis I disorder diagnosis other than Bipolar Disorder, including dementia, unstable medical illness or any contraindications to magnetic resonance imaging (MRI) will be excluded. Subjects may be concurrently prescribed other psychotropic medications, but dosages must be unchanged for one week prior to study entry and subjects must be willing to continue these medications during the study. All subjects must be able to provide written informed consent. Furthermore, subjects will be asked to complete a demographic information form.

Recruitment will take place through referrals from the McLean Hospital Geriatric Psychiatry Inpatient Service, Geriatric Psychiatry Outpatient Program: SAGE (Seniors Aging Gracefully Everyday) the Geriatric Psychiatry Outpatient Clinic, other inpatient, partial and outpatient psychiatric programs at McLean Hospital, the Cambridge Health Alliance, local geriatricians, the Harvard Division on Aging, local retirement communities, community psychiatrists, Partners Community Health Care PCP's, Massachusetts General Hospital and Brigham and Women's PCP network and similar external programs, as well as through radio and internet advertisements. We have obtained permission from the directors of both the Inpatient Service (Older Adult Unit) and Geriatric Psychiatry Outpatient Program (SAGE Program) to have a research assistant look through patient charts to identity eligible subjects. Once a potential subject has been identified, study staff will discuss the possibility of study participation with the patient's doctor to see if the study would be appropriate. If the doctor agrees about the patient's eligibility, the doctor will discuss the study with the patient and refer patients who are interested in participating to a member of our study staff.

Inclusion Criteria:

* 55 years or older
* Meet DSM-IV diagnostic criteria for Bipolar Disorder, Current Episode Depressed
* Montgomery Asberg Depression Rating Scale (MADRS) Score of >20
* If the MADRS score is <20 but >16, a diagnosis of bipolar disorder, current episode depressed, based on the Structured Clinical Interview of DSM IV TR (SCID) and Dr. Forester's initial interview would allow the subject to be included in the study.
* Young Mania Rating Scale (YMRS) Score of < 6
* If the YMRS score is >6 subjects can still be admitted if subjects do not meet clinical criteria for mania or hypomania at the time of screening
* Able to provide informed consent
* Must speak English
* Must be able to visit McLean Hospital for the screening visit and three-four study visits during the 4-5 week duration of the study
* Subjects may be taking other medications for bipolar depression including antidepressants, mood stabilizers and antipsychotic medications prior to Co-Q10 therapy, but will be encouraged not to have any dosage adjustments of these medications in the week before Co-Q10 is added and throughout their participation in the 4-week study. Changes to concomitant medication during the time between the screening and baseline visit or during the 4-week study due to a clinical need will be allowed. All concomitant medication changes will be noted in the study documents.

Exclusion Criteria (for bipolar disorder subjects and controls):

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder,
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, unipolar major depressive disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* History of drug hypersensitivity or intolerance to Coenzyme Q10.
* Current treatment with barbiturates.
* Benzodiazepines, and non-benzodiazepine sedative hypnotics (such as zolpidem (Ambien), may be used by subjects throughout the study as long as they are not taken within 12 hours of any MRI scan.
* Subjects diagnosed with a mitochondrial disorder.
* Subjects taking other putative mitochondrial enhancers (e.g., vitamin E, carnitine, creatine, Vitamin complex B, pramipexole) at the time of study entry.
* Subjects who either have metal objects in their bodies or work with metal or tools that could leave small pieces of metal in their eyes or skin will be excluded from the study as it is unsafe for them to have MRI scans.
* Women who are pregnant or are trying to become pregnant during their participation in the study.

Bipolar Subject Protocol

Summary:

This study is 4 weeks long, and will consist of 4 visits to the hospital. After an initial phone screening, subjects will come in for a baseline visit where they will meet with a psychiatrist to assess their past and current psychiatric and medical history. Subjects will also be administered the following mood rating scales: the MADRS (Montgomery-Asberg Depression Rating Scale), CGI (Clinical Global Impressions Scale), YMRS (Young Mania Rating Scale), GDS (Geriatric Depression Scale), and neuropsychological measures. If the subjects are fatigued, or if scheduling does not permit, screening procedures may be split into two visits that will occur within one week of each other. Within 7 days after the screening visit, subjects will come in for a baseline visit where they will have a 60 minute long 4.0T MRS scan. , The baseline and screening visit will take place before starting CoQ10. Subjects will be scheduled to have a 3T MRI scan for diagnostic purposes as soon as possible; however, this scan can take place at any point during the study. In addition, we will be obtaining a Magnetic Resonance Spectroscopy (MRS), functional Magnetic Resonance Imaging (fMRI) and a Diffusion Tensor Imaging study during the 3T MRI scan to obtain further information about specific nerve cell tracts or networks within the brain. During the fMRI portion of the scan we will not be asking you to perform any tasks; rather you will be asked to lay still with your eyes open and breathe normally. For all other portions of the scan there are no restrictions on closing your eyes. After the baseline visit, subjects will start taking CQ10 (dose schedule on page 13) for the next 4 weeks. Subjects will come in again at week 2 for a follow-up evaluation with Dr. Forester and will be administered the MADRS, CGI, and YMRS. At week 2, subjects will have another 4T scan, which will last 60 minutes. At week 4, subjects will have a third 60 minute long 4T MRI scan and will be re-administered the MADRS, CGI, YMRS, GDS and the neuropsychological tests (week 4 procedures may be split into two visits, within a week of each other, should subjects become fatigued, or if scheduling does not permit). The Wisconsin Card Sort Test and the Wechsler Test of Adult Reading (WTAR) will only be administered during the baseline visit and will not be administered to subjects during their last follow-up visits.

The study doctor will monitor response to treatment and changes in psychiatric clinical symptoms during the course of the 4 week treatment with CoQ10. If at any time during the study there are clinical changes that warrant a further clinical assessment by the study subject's primary clinician, the study principal investigator will refer the subject to their primary care clinician and/or psychiatrist as clinically needed.

Additionally, in the interest of having a standardized instrument to measure for side effects, we would like to include the Frequency and Intensity of Side Effects Ratings scale (FISER), a 3-item self-rated measure of medication side effects for our study. The principal investigator will continue to monitor for side effects during the clinical interview.

Control Subjects:

The control group will consist of 10 subjects (for the purposes of this study we would like to be able to recruit up to 30 subjects, with the goal of getting up to 10 to complete the protocol), ages 55-89, (matched with BPD group for age) without a known psychiatric disorder, unstable medical illness or any contraindications to MRI. A board certified geriatric psychiatrist will assess all control subjects for all current and past psychiatric disorders. Control subjects with any evidence of current or past psychiatric disorders will be excluded from the study. The Control Group will be recruited through contacts with the Harvard Division on Aging, local retirement communities and advertisements on the internet, in senior/city newspapers, and senior centers. Dr. Forester may also conduct in-service talks at local assisted living communities. Control subjects will meet the following conditions:

Inclusion Criteria:

* 55 years or older
* Able to provide informed consent
* Must speak English
* Women entering this study must be post-menopausal.

Exclusion Criteria:

Same criteria for the Bipolar Depressed group with the exception of the "first episode of mania" which is not applicable.

Control Subject Protocol

Control subjects (N=10) will be consented during the initial screening visit. The control subjects will not be given CoQ10. Otherwise, control subjects will follow the same protocol as the bipolar depressed subjects for the screening visit and will undergo the same psychiatric evaluation, implementation of rating scales and MRIs) as the bipolar depressed subjects (see above). The SCID and the clinical labs are not necessary components for the control protocol. Dr. Forester will assess current and past psychiatric symptoms and diagnoses with a standard clinical psychiatric interview. Approximately 1 week after the screening visit, control subjects will be scheduled to undergo the 4T MRS scan. The mood measures (MADRS and the YMRS) will be re-administered to the subjects during this visit. The 3T MRI scan will be scheduled as soon as possible but may be scheduled at any point during the subject's participation in the study. Control subjects will return 2 and 4 weeks after the baseline 4T visit to repeat the scan using the same protocol. Control subjects will have a total of three 4T MRS scans (during the baseline visit and the 2 and 4-week follow-up visits). The mood rating scales will be re-administered during the week 2 visit. Additionally, the mood measures and the neuropsychological tests will be re-administered during the week 4 visit. Control subjects will also be asked to complete a demographic information and clinical history form.

ELIGIBILITY:
Inclusion Criteria for Bipolar Depressed Subjects:

* 55 years or older
* Meet DSM-IV diagnostic criteria for Bipolar Disorder, Current Episode Depressed
* Montgomery Asberg Depression Rating Scale (MADRS) Score of >20
* If the MADRS score is <20 but >16, a diagnosis of bipolar disorder, current episode depressed, based on the Structured Clinical Interview of DSM IV TR (SCID) and Dr. Forester's initial interview would allow the subject to be included in the study.
* Young Mania Rating Scale (YMRS) Score of < 6
* If the YMRS score is >6 subjects can still be admitted if subjects do not meet clinical criteria for mania or hypomania at the time of screening
* Able to provide informed consent
* Must speak English
* Must be able to visit McLean Hospital for the screening visit and three-four study visits during the 4-5 week duration of the study
* Subjects may be taking other medications for bipolar depression including antidepressants, mood stabilizers and antipsychotic medications prior to Co-Q10 therapy, but will be encouraged not to have any dosage adjustments of these medications in the week before Co-Q10 is added and throughout their participation in the 4-week study. Changes to concomitant medication during the time between the screening and baseline visit or during the 4-week study due to a clinical need will be allowed. All concomitant medication changes will be noted in the study documents.

Exclusion Criteria for Bipolar Depressed Subjects:

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder,
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, unipolar major depressive disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* History of drug hypersensitivity or intolerance to Coenzyme Q10.
* Current treatment with barbiturates.
* Benzodiazepines, and non-benzodiazepine sedative hypnotics (such as zolpidem (Ambien), may be used by subjects throughout the study as long as they are not taken within 12 hours of any MRI scan.
* Subjects diagnosed with a mitochondrial disorder
* Subjects taking other putative mitochondrial enhancers (e.g., vitamin E, carnitine, creatine, Vitamin complex B, pramipexole) at the time of study entry.
* Subjects who either have metal objects in their bodies or work with metal or tools that could leave small pieces of metal in their eyes or skin will be excluded from the study as it is unsafe for them to have MRI scans.
* Women who are pregnant or are trying to become pregnant during their participation in the study.

Inclusion Criteria for Control Subjects:

* 55 years or older
* Able to provide informed consent
* Must speak English
* Women entering this study must be post-menopausal.

Exclusion Criteria for Control Subjects:

Same criteria for the Bipolar Depressed group with the exception of the "first episode of mania" which is not applicable, and patients with a lifetime history of substance dependence disorders, including alcohol, will be excluded.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bipolar subjects were recruited from the McLean Hospital Geriatric Psychiatry Inpatient and Outpatients services, and similar external programs, as well as through radio and internet advertisements. Controls through contacts with the Harvard Division on Aging, local retirement communities and advertisements on the internet, and senior centers.
Pre-assignment Details: Subjects who met DSM-IV diagnostic criteria for Bipolar Disorder and were currently depressed episode were assigned to the CoQ10 group. The CoQ10 group was to receive CoQ10 therapy for 4 weeks. Healthy control subjects no evidence of current or past psychiatric disorders were assigned to the Control group. This group did not receive CoQ10 therapy.
Groups:
- Control: Healthy controls with no evidence of current or past psychiatric disorders.
- CoQ10: Subjects with Bipolar disorder who received CoQ10 therapy for 4 weeks. Subjects in this group started at 400 mg of CoQ10 a day, and increased to 800 mg a day at 2 weeks.
Period: Overall Study
Arm/Group | Control | CoQ10
Started | 10 | 9
Completed | 6 | 8
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Screen Fail | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | CoQ10 | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (60.2) | 63 (50.05) | 62.21 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Concentrations of Cerebral Energetic Metabolites in Geriatric BPD and Older Controls at Baseline
Description: Tissue-specific (gray or white matter) concentrations of of Phosphocreatine (PCr), Beta-Nucleoside Triphosphate (bNTP), and Inorganic Phosphate (Pi) in geriatric BPD compared with healthy controls at baseline. Concentrations were measured using CSI P MRS scan at 4T. The analysis of signal intensity is done through integration of the area under the curve and is expressed in arbitrary units.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Integration Expressed as Arbitrary Unit
Arm/Group | Control | CoQ10
Number analyzed (Participants) | 6 | 8
Integration Expressed as Arbitrary Unit
  PCr in Gray Matter | 4.35 (0.16) | 3.94 (0.14)
  PCr in White Matter | 3.23 (0.15) | 3.06 (0.13)
  bNTP in Gray Matter | 2.63 (0.13) | 2.30 (0.12)
  bNTP in White Matter | 2.43 (0.12) | 2.38 (0.12)
  Pi in Gray Matter | 1.17 (0.06) | 1.39 (0.05)
  Pi in White Matter | 1.37 (0.04) | 1.23 (0.04)

2. Secondary Outcome: To Determine Effects of CoQ 10 on Bioenergetics (PCr and Beta NTP) in Older Adults With Bipolar Depression.
Description: Changes in Phosphocreatine and beta NTP (represented as adenosine triphosphate) in gray matter and white matter will be determined by measurements at Week 0 and Week 4 in Geri BD group challenged with CoQ10 and in healthy controls.
Time Frame: 4-week trial
Population: Healthy controls with no evidence of current or past psychiatric disorders, and subjects with Bipolar disorder who received CoQ10 therapy for 4 weeks. Subjects in the CoQ10 group started at 400 mg of CoQ10 a day, and increased to 800 mg a day at 2 weeks.
Measure: Least Squares Mean (Standard Error); unit: Integration Expressed as Arbitrary Unit
Groups:
- Control Baseline (Week 0): Healthy controls with no evidence of current or past psychiatric disorders.
- Control Week 4: Healthy controls with no evidence of current or past psychiatric disorders. Subjects did not receive study drug.
- CoQ10 Baseline (Week 0): Subjects with Bipolar disorder who had not yet received study drug.
- CoQ10 Week 4: Subjects with Bipolar disorder who received CoQ10 therapy for 4 weeks. Subjects in this group started at 400 mg of CoQ10 a day, and increased to 800 mg a day at 2 weeks.
Arm/Group | Control Baseline (Week 0) | Control Week 4 | CoQ10 Baseline (Week 0) | CoQ10 Week 4
Number analyzed (Participants) | 6 | 6 | 8 | 8
Integration Expressed as Arbitrary Unit
  Gray Matter Phosphocreatine | 4.350 (0.165) | 4.425 (0.168) | 3.944 (0.143) | 4.435 (0.151)
  White Matter Phosphocreatine | 3.226 (0.150) | 3.424 (0.151) | 3.063 (0.127) | 2.997 (0.132)
  Gray Matter Adenosine Triphosphate | 2.620 (0.130) | 2.649 (0.133) | 2.283 (0.113) | 2.088 (0.117)
  White Matter Adenosine Triphosphate | 2.417 (0.120) | 2.148 (0.121) | 2.376 (0.102) | 2.844 (0.105)

ADVERSE EVENTS:
Arm/Group | Control | CoQ10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | CoQ10 (N=9)
Difficulty Sleeping (General disorders) | 0 (0) | 1 (1)
Mild Nausea (General disorders) | 0 (0) | 1 (1)
Discomfort in MRI (General disorders) | 1 (1) | 0 (0)
Reduced Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No